CLINICAL TRIAL: NCT00981591
Title: A Randomized, Double Blind, Placebo-controlled Pilot Study of the Safety and Effective Dosing of Inhaled Iloprost in Pediatric Patients With Pulmonary Hypertension Treated With Inhaled Nitric Oxide
Brief Title: Inhaled Iloprost as an Adjunct to Inhaled Nitric Oxide in Pediatric Critical Care Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No patients recruited
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Actelion (Industry)
Responsible Party: Principal Investigator, Delphine Yung, Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCIL-001-12806
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Pulmonary Hypertension; Neonatal Hypoxic Respiratory Failure; Persistent Pulmonary Hypertension of Newborn; Congenital Heart Defects; Acute Respiratory Distress Syndrome
Keywords: Iloprost; Nitric oxide; Mechanical ventilator
MeSH Terms: conditions — Hypertension, Pulmonary; Persistent Fetal Circulation Syndrome; Heart Defects, Congenital; Respiratory Distress Syndrome | interventions — Iloprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Iloprost (Experimental)
  Interventions: Drug: Iloprost
- Inhaled Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iloprost — Inhaled via Aerogen nebulizer, 0.5 mcg/kg every 2 hours; uptitrated to effect, to maximum dose of 30 mcg every 30 minutes
  Other Names: Ventavis
  Arms: Inhaled Iloprost
Drug: Placebo — Inhaled via Aerogen nebulizer, 0.5 mcg/kg every 2 hours or more
  Arms: Inhaled Placebo

SUMMARY:
The purpose of this study is to determine whether inhaled iloprost is safe and effective in pediatric patients with pulmonary hypertension who are sick in the intensive care unit.

DETAILED DESCRIPTION:
Inhaled nitric oxide (NO) is used in the management of all causes of pediatric pulmonary hypertension. Despite widespread use of nitric oxide to treat critically ill mechanically-ventilated pediatric patients with pulmonary hypertension, response to therapy is not universal. Nitric oxide fails to improve oxygenation in approximately 30% of these patients. Nonresponders to nitric oxide have few treatment options. Iloprost is the only other medication approved for inhalational delivery in the treatment of pulmonary hypertension. Inhalation therapy for pulmonary vasodilatation in critically ill children is inherently more attractive than oral or intravenous therapies due to the ability to deliver medication directly to the lung and to decrease systemic effects. The use of inhaled iloprost has been reported to decrease pulmonary vascular resistance in many pediatric pathologic settings, including combination therapy with nitric oxide.

ELIGIBILITY:
Inclusion Criteria:

* Birth to 21 years of age
* Diagnosis of pulmonary hypertension must fit into one of three categories

  * neonatal hypoxic respiratory failure
  * congenital heart disease
  * acquired/acute respiratory distress syndrome (lung disease)
* Parents of subject must be able and willing to give written informed consent and comply with the requirements of the study protocol and must authorize release and use of protected health information
* Patients who remain on nitric oxide at 12 to 18 hours after initiation
* Patients who are transferred to an intensive care unit already on inhaled nitric oxide from another institution will be treated as if nitric oxide therapy was started at the time of admission to the unit
* Patients will be enrolled only after a clinical decision to treat with nitric oxide has been made by the treating physician

Exclusion Criteria:

* Corrected gestational age less than 35 weeks
* Patients with potentially fatal non-cardiopulmonary co-morbidities (e.g. hepatic, neurologic, renal)
* Known or suspected fatal genetic syndrome
* Patient with cardiac failure secondary to significant left-sided obstructive lesions
* Patient on ECMO
* Patient on any other form of prostacyclin
* Patient on any medication with known NO production, e.g., nitroprusside
* Patient on an endothelin receptor antagonist (e.g. bosentan)
* Patient on sildenafil
* Patient on whom clinicians do not agree to follow standard inhaled nitric oxide weaning protocol
* Patients who have known hypersensitivity to prostacyclin or any of its components
* Patient who is pregnant
* Patient with platelet count less than 50,000

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To determine the safety and effective dosing of inhaled iloprost in mechanically ventilated pediatric patients with pulmonary hypertension. | For the duration of time that the subject is receiving the study drug

SECONDARY OUTCOMES:
Time to wean off iNO. | When the participant is successfully weaned off study drug
Time to extubation. | When the participant is successfully weaned off study drug
Total cost of iNO. | When the participant is successfully weaned off study drug
Incidence of rebound phenomenon, as defined by the need to return to a higher iNO dose after a previous wean. | When the participant is successfully weaned off study drug
Time to ICU discharge | When the participant is successfully weaned off study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Yung, MD, Principal Investigator — Seattle Children's Hospital